CLINICAL TRIAL: NCT01299870
Title: Keishibukuryogan (Japanese Herbal Supplement) for the Adjunctive Treatment of Catamenial Epilepsy in Adult: Safety Study
Brief Title: Catamenial Epilepsy Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Timothy Welty, PharmD (Other)
Responsible Party: Sponsor-Investigator, Timothy Welty, PharmD, Professor and Chair of Pharmacy Practice, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12416
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — keishibukuryogan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AED treatment plus placebo (Active Comparator)
  Interventions: Drug: AED treatment plus placebo
- Keishibukuryogan (Experimental)
  Interventions: Drug: Keishibukuryogan

INTERVENTIONS:
Drug: AED treatment plus placebo — Your usual AED(s) treatment with placebo for 12 weeks followed by 4 weeks washout period, and then Keishibukuryogan, (2.5 g of granulate filled in capsules) three times a day for a total of 7.5 g a day with your usual AED(s) treatment for 12 weeks.
  Arms: AED treatment plus placebo
Drug: Keishibukuryogan — Keishibukuryogan, (2.5 g of granulate filled in capsules) three times a day for a total of 7.5 g a day with your usual AED(s) for 12 weeks followed by 4 weeks washout period, and then your usual AED(s) treatment with placebo for 12 weeks.
  Arms: Keishibukuryogan

SUMMARY:
Epilepsy is a disorder in the brain. The brain is full of "nerve" cells. Nerve cells have normal electrical activity to control the many functions of the body. Sometimes nerve cells do not function normally due to many different reasons such as disease, an injury or because the brain didn't develop normally at birth. When nerve cells do not function normally the electrical activity that controls things like muscles and body movement can get mixed up and cause seizures. When a seizure occurs, sometimes a person loses control of body movement, and/or bodily functions. When a seizure occurs, a person may become unconscious, and/or senses may be affected. Seizures can occur at any time, without warning, and can lead to many health problems.

"Catamenial epilepsy" is specific form of epilepsy in women. It is closely related to the menstrual cycle. In this form of epilepsy seizures increase around the menstrual period.

By doing this study, researchers hope to learn whether Keishibukuryogan add-on therapy with antiepileptic drugs is safe for women with epilepsy.

DETAILED DESCRIPTION:
It is known that the female hormone levels in epilepsy patients are different from healthy women. These hormonal differences may be part of the cause of catamenial epilepsy. It is estimated that at least 1 in every 3 women with epilepsy have catamenial epilepsy. Although many antiepileptic drugs are available, it is very difficult to control these seizures. In the past, studies using antiepileptic drugs and hormonal agents were done to treat catamenial epilepsy. However, those medications did not work well and caused side effects.

Keishibukuryogan is a traditional Japanese herbal medication. It is made of 5 natural herbs (cinnamon bark, hoelen, moutan bark, peony root, and peach kernel). It is used to treat disorders in women like menopause and menstrual cycle problems. This is the first study to examine the safety of Keishibukuryogan in women with epilepsy. As such, Keishibukuryogan and your current antiepileptic drug(s) will be given to you during the study.

Keishibukuryogan is a dietary supplement in the United States. It can be bought without a prescription. The safety and efficacy of Keishibukuryogan has not been studied in epilepsy. However, it has been used safely in Japan and other Asian countries for years.

ELIGIBILITY:
Inclusion Criteria

1. Female with a positive diagnosis of epilepsy, and
2. Women with epilepsy (WWE) patients who have seizures and treated with AEDs and no dosage changes in the past 30 days, and
3. WWE patients with regular menstrual period with range of 28 ± 7 days.
4. WWE patients with age range between 21 and 45 years old.
5. WWE patients who are willing and able to give signed informed consent form are eligible to participate in this study.
6. WWE who agree to use non-hormonal forms of contraception for the duration of this study.

   No hormonal Intra-Uterine Device is allowed for the duration of this study.
7. Patients with a history of cancer must be in remission for at least 5 years.

Exclusion Criteria

1. History of status epilepticus in the last 12 months
2. Current diagnosis of polycystic ovary syndrome and/or endometriosis
3. Pregnant or breast feeding
4. Allergy to any ingredients in KBG (cinnamon, hoelen, moutan bark, peony root, or peach kernel)
5. Patients who are receiving warfarin and/or antiplatelet drugs
6. Severe cardiovascular, renal or hepatic impairment (i.e., coronary heart disease, myocardial infarction, renal failure, hepatitis) or history of those diseases
7. Any other unstable diseases (e.g., mental disease, infection, cancer)
8. Lab values at screening phase showing 1.5 times above the upper range of normal
9. Patients who are receiving phenytoin will be excluded (since a potential interaction between phenytoin and peony root was reported)

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To determine if Keishibukuryogan is safe for WWE | up to 36 weeks
  Keishibukuryogan is commonly used in Japan, but has not been formally studied in people with epilepsy. This study is designed to determine if KBG is safe to use in women with epilepsy (no increase of seizure and no adverse reactions).

SECONDARY OUTCOMES:
To determine if KBG changes seizure frequency in WWE, with a focus on increases in seizure frequency. | up to 36 weeks
  Based on the basic animal data, KBG has antiepileptic properties and may be beneficial for WWE.
To determine if KBG alters progesterone levels in WWE. | up to 36 weeks
  Based on the basic animal data, KBG altered serum progesterone level. Therefore, we would like to examine how KBG affects serum progesterone level.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Welty, Pharm D, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States